CLINICAL TRIAL: NCT02806635
Title: Web-based Marriage Preparation/Enrichment and Divorce Prevention for Low-Income Couples
Brief Title: Web-based Programs to Improve and Strengthen Romantic Relationships
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Children's Bureau - Administration for Children and Families (Other)
Responsible Party: Principal Investigator, Brian D Doss, Ph.D., Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20160451
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Romantic Relationship
Keywords: Relationship Distress; Relationship Satisfaction; Marriage; Web-based; Internet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Waitlist (No Intervention): Participants are assessed start, during, and end wait list; however, no active intervention is given.
- OurRelationship (Experimental): The OurRelationship program is based on Integrative Behavioral Couple Therapy and encourages couples to select, understand, and solve a relationship problem. Partners complete the majority of the web-based program on their own and come together for three key conversations with their partner. The first conversation between partners centers on discussing possible core relationship issues and jointly deciding on the problem(s) to focus on during the program. During the second conversation, both partners' previous written responses are displayed on the screen and conversation is encouraged. During the final conversation, couples share their strategies to decrease stress, improve patterns of communication, and engage in problem-solving exercises specific to their core issue(s).
  Interventions: Behavioral: OurRelationship
- PREP Online (Experimental): The PREP Online program is based on the in-person Prevention and Relationship Enhancement Program. The PREP Online program consists of seven sections of material. In each section, new information and skills are presented, videos demonstrate real couples practicing the skills, participants are encouraged to discuss the information in the context of their own relationship, and a multiple choice quiz reiterates and summarizes the section. In addition to the core educational materials, couples are asked to complete six additional online and offline homework assignments (one per week), each lasting approximately one hour.
  Interventions: Behavioral: PREP Online

INTERVENTIONS:
Behavioral: OurRelationship
  Other Names: Integrative Behavioral Couple Therapy
  Arms: OurRelationship
Behavioral: PREP Online
  Other Names: Prevention and Relationship Enhancement
  Arms: PREP Online

SUMMARY:
This study investigates the effectiveness of www.OurRelationship.com, which provides self-help, web-based programs to improve romantic relationships and related outcomes. Couples will be randomly assigned to complete the OurRelationship program, the PREP Online program, or a wait-list control group and followed for six months.

DETAILED DESCRIPTION:
Nationwide, lower-income (LI) couples (those with household incomes <200% of the federal poverty level) - many of whom are also African American, Hispanic/Latino, or rural couples - face numerous challenges to their relationships. Chief amongst those challenges are: 1) higher risk of relationship problems and 2) lack of access to effective relationship services to prevent or intervene with relationship distress. Compared to higher-income couples, LI married and cohabiting couples are significantly more likely to divorce or separate and report lower relationship quality. Unfortunately, LI couples are least likely to receive interventions to prevent or solve relationship problems. To overcome these barriers, we propose to test the effectiveness of two effective web-based curricula - OurRelationship and PREP Online.

A total of 750 LI couples will be recruited nationwide and randomly assigned to the PREP Online program, the OurRelationship program, or a wait-list control group and followed for six months. Once randomly assigned to group, couples will be assessed at one month, two months, four months, and six months following randomization. After couples randomized to the wait-list control group finish their waiting period, they will be able to select the program they would like to complete (OurRelationship or ePREP) but will not complete research assessments during or following their participation in the program. Interested couples can find out more information (and sign up for the study) at www.OurRelationship.com

ELIGIBILITY:
Inclusion Criteria:

1. They are married, engaged, or have been cohabiting with their partner for at least six months
2. They are both located in the United States
3. Both partners are willing to participate in the study
4. Both partners are between the ages of 18 and 64 (inclusive)
5. Both partners are fluent readers of the English language (as the program materials are currently only available in English).
6. Couples report a household income at or below 200% of the Federal Poverty Level.

Exclusion Criteria:

1. Severe domestic violence
2. Inadequate internet connection
3. Previous participation in OR, PREP-O, in-person PREP, or its variants
4. Current participation in other relationship programs
5. Current participation in an evaluation funded by Administration for Children and Families

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1484 (Actual)
Dates: Start 2016-10-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Relationship Satisfaction | Baseline and 6 months
  Four-item Couple Satisfaction Index (CSI) self-report measure

SECONDARY OUTCOMES:
Change in Relationship Knowledge | Baseline and 6 months
  Six-item, self-report measure of relationship knowledge
Change in Communication Skills | Baseline and 6 months
  Seven-item, self-report measure of communication skills

CONTACTS AND LOCATIONS:
Overall Officials: Brian Doss, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be provided to Administration for Children and Families to facilitate secondary data analyses.

REFERENCES:
- [Derived] Doss BD, Knopp K, Roddy MK, Rothman K, Hatch SG, Rhoades GK. Online programs improve relationship functioning for distressed low-income couples: Results from a nationwide randomized controlled trial. J Consult Clin Psychol. 2020 Apr;88(4):283-294. doi: 10.1037/ccp0000479. PMID 32134290